CLINICAL TRIAL: NCT02905747
Title: The Effect of Medical Exercise Therapy on Pain, Function and Physical Activity in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/872
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Exercise Therapy; Musculoskeletal Pain; Knee osteoarthritis; Physical Therapy Modalities
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Exercise Therapy (Experimental): Medical Exercise Therapy (MET) developed by Oddvar Holten
  Interventions: Behavioral: Medical Exercise Therapy

INTERVENTIONS:
Behavioral: Medical Exercise Therapy — physiotherapy intervention with Medical exercise therapy (MET) during 3 months

SUMMARY:
The aim of the project is to investigate effects of medical exercise therapy (MET) on patients with knee osteoarthritis. MET is a common physical therapy intervention, and the project aim to strengthen the evidence of this intervention. An experimental cohort design is chosen, and 20 participants will be followed for 6 months. Assessments will be clinical tests, questionnaires and accelerometer measurements before, during, and after a 3 month period of exercise (3 days per week) with a physical therapist. The project will answer if a 3 month physical therapy intervention using MET causes changes in pain level, function and activity level for patients with knee osteoarthritis. In addition, it will investigate whether a single global endurance workout for 30 minutes will have an effect on pain level for these patients

ELIGIBILITY:
Inclusion Criteria:

* x-ray verified knee osteoarthritis (Kellegren & Lawrence grade I-III)
* Loss of function and withstanding pain >3 months

Exclusion Criteria:

* physical therapy treatment during the last 3 months
* knee injury
* inflammatory arthritis
* symptoms from the hip joints greater than the knee pain
* planned knee surgery the next 6 months
* heart and lung disorders or other health issues affecting the ability to complete the intervention

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
pain | 6 months
  visual analog scale
Activity level | 6 months
  Accelerometer
Function | 6 months
  30 second chair stand test

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Østerås, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Osteras H, Paulsberg F. The Effect of Medical Exercise Therapy on Pressure Sensitivity in Patients with Knee Osteoarthritis: A Cohort Pilot Study. Pain Ther. 2019 Jun;8(1):79-87. doi: 10.1007/s40122-019-0121-5. Epub 2019 Mar 30. PMID 30929225